CLINICAL TRIAL: NCT02109042
Title: A Multiple Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Blosozumab Proposed Phase 3 Formulation in Postmenopausal Women
Brief Title: A Study of Blosozumab (LY2541546) in Postmenopausal Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15172; I2M-MC-GSDM (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2017-09

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — blosozumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blosozumab (Experimental): Weekly SC injections of blosozumab for 6 weeks.
  Interventions: Drug: Blosozumab

INTERVENTIONS:
Drug: Blosozumab — Administered subcutaneously
  Other Names: LY2541546

SUMMARY:
The purpose(s) of this study is to measure how much of the study drug gets into the blood stream and how long it takes the body to get rid of it when given in multiple doses, subcutaneously (SC) (by inserting a needle just under the surface of the skin in the lower abdominal area), to postmenopausal (PMP) female participants. Information about any side effects that may occur will also be collected.

This study will also be looking for special markers called "biomarkers" that can be used to study osteoporosis and/or the effects of the study drug.

There will be 2 parts to this study. The first part will last approximately 6 weeks and the second part will last approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Part A: Overtly healthy PMP females
* Part B: PMP women who are currently taking oral bisphosphonates
* Have a body mass index (BMI) at screening of 19.0 to 35.0 kilogram per square meter (kg/m^2)

Exclusion Criteria:

* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Have known allergies to blosozumab, its constituents, or related compounds
* Have an abnormality in the 12-lead electrocardiogram (ECG)

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Weekly Subcutaneous Blosozumab Injections: Blosozumab was to be administered as a subcutaneous (SC) injection (90 milligrams per milliliter (mg/mL) solution in prefilled syringes) weekly for 6 weeks.
  A 180 mg loading dose (2 × 1 mL injections) was administered on Day 1 of Week 1 followed by 5 planned once weekly 90 mg doses (single 1 mL injection) beginning on Day 1 of Week 2.
Period: Overall Study
Arm/Group | Weekly Subcutaneous Blosozumab Injections
Started | 15
Received at Least 1 Dose of Study Drug | 15
Received 180 mg Loading Dose | 15
Receive at Least 1 Subsequent 90 mg Dose | 15
Completed | 0
Not Completed | 15
Not completed — Sponsor Decision | 15

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 SC Blosozumab injection.
Groups:
- Weekly SC Blosozumab Injections: Blosozumab was to be administered as a SC injection (90 mg/mL solution in prefilled syringes) weekly for 6 weeks.
  A 180 mg loading dose (2 × 1 mL injections) was administered on Day 1 of Week 1 followed by 5 planned once weekly 90 mg doses (single 1 mL injection) beginning on Day 1 of Week 2.
Arm/Group | Weekly SC Blosozumab Injections
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Blosozumab
Description: The mean maximum observed drug concentration of Blosozumab during 1 dosing interval was reported.
Time Frame: Predose and daily up through 7 days postdose
Population: Participants who received at least 1 SC Blosozumab injection and had evaluable PK concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles per milliliter
Arm/Group | Weekly SC Blosozumab Injections
Number analyzed (Participants) | 15
picomoles per milliliter | 59.8 (54)

2. Primary Outcome: PK: Area Under the Concentration Curve of Blosozumab
Description: The mean area under the concentration of Blosozumab versus time curve during 1 dosing interval was reported.
Time Frame: Predose and daily up through 7 days postdose
Population: Participants who received at least 1 SC Blosozumab injection and had evaluable PK concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles times hours per milliliter
Arm/Group | Weekly SC Blosozumab Injections
Number analyzed (Participants) | 15
picomoles times hours per milliliter | 7160 (58)

ADVERSE EVENTS:
Groups:
- 180 mg SC Blosozumab Injection: Blosozumab was planned to be administered as a SC injection (90 mg/mL solution in prefilled syringes) weekly for 6 weeks.
  A 180 mg loading dose (2 × 1 mL injections) was administered on Day 1 of Week 1.
- 90 mg SC Blosozumab Injections: Blosozumab was planned to be administered as a SC injection (90 mg/mL solution in prefilled syringes) weekly for 6 weeks.
  Once weekly 90 mg dose (single 1 mL injection) were administered beginning on Day 1 of Week 2.
  Data from all participants who received at least 1 90 mg/mL SC Blozozumab injection are included.
Arm/Group | 180 mg SC Blosozumab Injection | 90 mg SC Blosozumab Injections
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 14/15 | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 180 mg SC Blosozumab Injection (N=15) | 90 mg SC Blosozumab Injections (N=15)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Injection site dermatitis (General disorders) | 0 (0) | 5 (5)
Injection site erythema (General disorders) | 11 (20) | 13 (26)
Injection site haemorrhage (General disorders) | 3 (3) | 2 (2)
Injection site hypersensitivity (General disorders) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 2 (2)
Injection site oedema (General disorders) | 9 (15) | 4 (4)
Injection site pain (General disorders) | 3 (6) | 6 (10)
Injection site pruritus (General disorders) | 0 (0) | 8 (13)
Injection site swelling (General disorders) | 0 (0) | 4 (4)
Malaise (General disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Before Part B of the study, Eli Lilly and Company decided to stop any further dose administration; no participants entered Part B of the study. The decision was not based on safety concerns, but rather tolerability issues (injection site reactions).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days